CLINICAL TRIAL: NCT03679065
Title: Prophylactic Paracetamol or Dexamethasone for Post-spinal Anesthesia Shivering in Patients Undergoing Non-obstetric Surgeries: a Randomized Controlled Trial
Brief Title: Prophylactic Paracetamol or Dexamethasone for Post-spinal Anesthesia Shivering
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Dr.Ibrahim Mamdouh Esmat, Assistant Professor, M.D., Department of Anesthesia and Intensive Care, Ain- shams University, Egypt., Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: R 49 / 2018
Record Dates: First submitted 2018-09-19; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Shivering
MeSH Terms: interventions — Acetaminophen; Dexamethasone; dexamethasone 21-phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- P (Paracetamol) group:(n=100) (Active Comparator)
  Interventions: Drug: Paracetamol
- D (Dexamethasone) (Dex) group: (n=100) (Active Comparator)
  Interventions: Drug: Dexamethasone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Each patient received 1g paracetamol tablet orally with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 minutes as a placebo for Dex solution 2 hours preoperatively.
  Arms: P (Paracetamol) group:(n=100)
Drug: Dexamethasone — Each patient received a placebo tablet identical to paracetamol tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 minutes, 2 hours preoperatively.
  Other Names: Dexamethasone phosphate
  Arms: D (Dexamethasone) (Dex) group: (n=100)
Drug: Placebo — Each patient received a placebo tablet identical to paracetamol tablet orally with sips of water and 100 ml 0.9% NS IVI over 15 minutes as a placebo for Dex solution 2 hours preoperatively.
  Arms: Placebo

SUMMARY:
This study was conducted to evaluate the effects of a prophylactic dose of oral paracetamol on shivering compared with prophylactic intravenous infusion (IVI) dexamethasone in patients undergoing non-obstetric surgeries under spinal anesthesia.

DETAILED DESCRIPTION:
Enrollment After approval by the institute ethics committee, this study was conducted at Ain-Shams university hospitals, from the1st of March 2018 till the 31st of August 2018, on 300 patients aged 18-60 years and body weight 60-100 Kg of the American Society of Anesthesiologists (ASA) physical status I or II who underwent non-obstetric surgeries under spinal anesthesia were enrolled in this study.

Patient's refusal, duration of surgery more than 120 min, obesity with body mass index (BMI) >35 kg/m2, generalized infection or localized infection at level of blockade, neurologic disease, coagulation disorder, patients with hypo- or hyperthyroidism, cardiopulmonary disease, psychological disorders, a need for blood transfusion during surgery, an initial body temperature >38.0C or <36.0C, a known history of alcohol or substance abuse, or receiving vasodilators, or medications likely to alter thermoregulation excluded the patient. from the study Randomization and Blinding This study was designed to be a randomized, placebo-controlled, double-blinded parallel study. Following enrollment, patients were randomized into 3 equal groups;

1. The P (Paracetamol) group:(n=100) each patient received 1g paracetamol tablet orally with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 minutes as a placebo for Dex solution 2 hours preoperatively.
2. The D (Dexamethasone) group: (n=100) each patient received a placebo tablet identical to paracetamol tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 minutes, 2 hours preoperatively.
3. The C (Control) group: (n=100) each patient received a placebo tablet identical to paracetamol tablet orally with sips of water and 100 ml 0.9% NS IVI over 15 minutes as a placebo for Dex solution 2 hours preoperatively.

Randomization was done using computer-generated table of random numbers in a 1:1 ratio in opaque and sealed envelope (SNOSE). The assigned treatment was written on a card and sealed in opaque envelopes consecutively numbered. These envelopes were opened just immediately before infusing the medication in the patient's room. The study drugs were prepared by the hospital pharmacy and follow-up of patients were conducted by anesthesia residents not involved in any other part of the study.

Study Protocol On arrival in the operating theatre, all patients had an inserted venous cannula. I.V. fluids were preheated to 37oC. No other warming device was used. Lactated Ringer's solution was warmed to 37 oC and was infused at 10 ml/kg over 30 min before spinal anesthesia. The infusion rate was reduced to 6 ml/ kg.

Subarachnoid anesthesia was instituted at either L3/4 or L4/5 interspaces. Hyperbaric bupivacaine, 5 mg /ml, 15 mg was injected using a 25 G Quincke spinal needle.

Supplemental oxygen (5 liter/ min) was delivered via a facemask during the operation. All patients were covered with one layer of surgical drapes over the chest, thighs, and calves during the operation and one cotton blanket over the entire body after operation. The operating and recovery rooms temperatures were maintained at 23-25°C with approximately 60% humidity.

Assessment parameters Heart rate, mean arterial pressure (MAP), and peripheral oxygen saturation were recorded using standard noninvasive monitors before intrathecal injection and thereafter at 5, 10, 15, 20 minutes then every 10 minutes to complete 90 minutes from the intrathecal injection.

Sensory levels were assessed by pinprick to determine the peak sensory level and time to two segment regression in minutes. Motor block was assessed by using Modified Bromage scale(16) (0 = no block 1 = hip block, 2 = hip and knee block, 3 = hip, knee, and ankle block) to determine the time to reach complete motor block and duration of motor blockade (minutes).

Sedation score was assessed with a four-point scale as per Filos et al.(17): 1: Awake and alert. 2: Somnolent, but responsive to verbal stimuli. 3: Somnolent, arousable to physical stimuli. 4: Unarousable.

Body temperature (axillary temperature) was recorded with an axillary thermometer. The ambient temperature was measured by a wall thermometer. The ambient temperature was maintained at 25oC with constant humidity.

Shivering if occurred was graded using a scale similar to that validated by Badjatia et al (18):

1. None: no shivering noted on palpation of the masseter, neck, or chest wall
2. Mild: shivering localized to the neck and/or thorax only
3. Moderate: shivering involved gross movement of the upper extremities (in addition to neck and thorax)
4. Severe: shivering involved gross movements of the trunk and upper and lower extremities.

Shivering was assessed immediately before the block and every 10 minutes till the end of surgery and for another 20 min in the recovery room. Grade 3 or 4 of shivering score was regarded failure of prophylaxis, meperidine 25 mg IV was administered and no assessment of shivering was done.

Side-effects, including hypotension (defined as a decrease in MAP of more than 20% from baseline or a decrease of arterial blood pressure below 90 mmHg and baseline MAP was calculated from three measurements taken on the ward before surgery) was treated by crystalloid infusion and if necessary ephedrine 5 mg IV was administered. The amount of ephedrine given in each group was recorded. Bradycardia was considered if the heart rate <50 beats/min and was treated with IV atropine (0.01mg/kg). If there was respiratory depression (RR < 12 bpm) and a decrease in arterial SpO2 (<90%), it was treated with oxygen through a transparent face mask. Incidence of nausea and vomiting during early 2 hours postoperatively were recorded. IV granisetron (1 mg) was given in case of vomiting or after 2 successive episodes of nausea.

Patient's satisfaction was done by asking the patient to answer the question, "How would you rate your experience after the surgery?" using a 7-point Likert verbal rating scale(19): [Figure 1] and acceptable satisfaction score of the patient being 5-7.

Likert scale:

1 2 3 4 5 6 7 Extremely dissatisfied Dissatisfied Somewhat dissatisfied Undecided Somewhat satisfied Satisfied Extremely satisfied Figure 1: A 7-point Likert-like verbal rating scale for assessment of patients' satisfaction(19).

Endpoint: The study end point was 20 minutes after the end of the procedure (in the recovery room)

Primary Outcome Measure:

Total participants received pethidine for treatment of post-spinal shivering in the three groups till 20 minutes after the end of the procedure (in the recovery room)

Secondary Outcome Measures:

* Incidence, onset, severity and duration of post-spinal shivering.
* Time to first analgesic request, from the end of surgery up to approximately six hours after surgery
* Incidence of hypotension.
* Incidence of bradycardia.
* Incidence of nausea and vomiting during early 2 hours postoperatively.
* Patient' satisfaction towards shivering prophylaxis was assessed 24 hours after the procedure.

  3-Analysis of Data:

Depending on Gholami et al., 2016 who found that shivering was 18% and 64.0% in paracetamol and control respectively(20) and on El Bakry et al., 2016 who found that shivering was 20.0% and 50.0% in dexamethasone and control respectively(21) and assuming the power= 0.80 and α=0.05, and by using PASS 11th release the minimal sample size for an equal controlled study to detect a significant statistical difference between paracetamol & dexamethasone and control was 80 women in each group. We recruited 100 women in each group for possible attrition(22).

The collected data were coded, tabulated, and statistically analyzed using IBM SPSS statistics (Statistical Package for Social Sciences) software version 22.0, IBM Corp., Chicago, USA, 2013.

ELIGIBILITY:
Inclusion Criteria:

* • on 300 patients aged 18-60 years

  * of the American Society of Anesthesiologists (ASA) physical status I or II
  * underwent non-obstetric surgeries under spinal anesthesia. A written informed consent was obtained from all patients to participate in the study.

Exclusion Criteria:

* • Patient's refusal,

  * duration of surgery more than 120 min,
  * obesity with body mass index (BMI) >35 kg/m2,
  * generalized infection or localized infection at level of blockade,
  * neurologic disease,
  * coagulation disorder,
  * patients with hypo- or hyperthyroidism,
  * cardiopulmonary disease,
  * psychological disorders,
  * a need for blood transfusion during surgery,
  * an initial body temperature >38.0C or <36.0C,
  * a known history of alcohol or substance abuse,
  * or receiving vasodilators, or medications likely to alter thermoregulation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Total participants received pethidine for treatment of post-spinal shivering in the three groups till 20 minutes after the end of the procedure (in the recovery room) | Till 20 minutes after the end of the procedure (in the recovery room)
  Total participants received pethidine for treatment of post-spinal shivering in the three groups till 20 minutes after the end of the procedure (in the recovery room)

CONTACTS AND LOCATIONS:
Locations (1):
- Ibrahim Mamdouh Esmat, Heliopolis, Cairo Governorate, Egypt

REFERENCES:
- [Derived] Esmat IM, Mohamed MM, Abdelaal WA, El-Hariri HM, Ashoor TM. Postspinal anesthesia shivering in lower abdominal and lower limb surgeries: a randomized controlled comparison between paracetamol and dexamethasone. BMC Anesthesiol. 2021 Oct 30;21(1):262. doi: 10.1186/s12871-021-01483-7. PMID 34717535